CLINICAL TRIAL: NCT06946121
Title: Comparison Between the Intrauterine Lidocaine and Warm Saline Distention Medium for Pain Relief During Office Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 364
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine group (Experimental): 50 women undergoing diagnostic outpatient office hysteroscopy proceeded by infusions of intrauterine lidocaine 2% and normal saline at room temperature.
  Interventions: Drug: Lignocaine
- Saline group (Placebo Comparator): 50 women undergoing diagnostic outpatient office hysteroscopy using warmed normal saline distention medium
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lignocaine — 50 women undergoing diagnostic outpatient office hysteroscopy proceeded by infusions of intrauterine lidocaine 2% and normal saline at room temperature.
  Arms: Lignocaine group
Drug: Saline — 50 women undergoing diagnostic outpatient office hysteroscopy using warmed normal saline distention medium.
  Arms: Saline group

SUMMARY:
Procedure:

The procedure was done in the lithotomy position during the postmenstrual period.

We used a 30° angle 2.9 mm rigid hysteroscopy with 3.8 mm diagnostic sheath [TEKNO®, LIGHT XA 180, Germany].

Vaginoscopic approach was used for insertion of the hysteroscopy in all cases (no use of speculum or tenaculum).

The hysteroscopy was gently introduced into the uterine cavity after visualization of the cervix and identification of the external os.

We used saline as the distension medium and the maximum pressure was set at 70 to 80 mm Hg by an automated hysteroscopic pump system (Hysteromat II, Karl Storz), which automatically measured intrauterine fluid pressure. In lidocaine group: we added 5 ml of lidocaine 2% to 500 ml of saline solution that was used as a distention medium.

The uterine cavity and tubal ostia were systematically visualized. All procedures were done by an operator using the same equipment.

DETAILED DESCRIPTION:
A written consent was taken from eligible women on admission after explaining the aim of the research, procedure, expected value, outcome, and possible adverse effects, with full details provided to them. They were informed that their participation in this study is voluntary and they may refuse to participate or withdraw from the study at any time.

After fulfilling inclusion and exclusion criteria, patients were equally randomized by simple randomization with a 1:1 allocation ratio into two groups using computer-generated random numbers. The envelopes were kept in the office hysteroscopy room in a closed box. Each of the envelopes was taken out of the box sequentially according to the order of women attendance.

Procedure:

The procedure was done in the lithotomy position during the postmenstrual period.

We used a 30° angle 2.9 mm rigid hysteroscopy with 3.8 mm diagnostic sheath [TEKNO®, LIGHT XA 180, Germany].

Vaginoscopic approach was used for insertion of the hysteroscopy in all cases (no use of speculum or tenaculum).

The hysteroscopy was gently introduced into the uterine cavity after visualization of the cervix and identification of the external os.

We used saline as the distension medium and the maximum pressure was set at 70 to 80 mm Hg by an automated hysteroscopic pump system (Hysteromat II, Karl Storz), which automatically measured intrauterine fluid pressure. In lidocaine group: we added 5 ml of lidocaine 2% to 500 ml of saline solution that was used as a distention medium.

The uterine cavity and tubal ostia were systematically visualized. All procedures were done by an operator using the same equipment.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old.

Indications of diagnostic office hysteroscopy as:

Suspicion of the intracavitary lesion. Abnormal uterine bleeding. Abnormal endometrial thickening. Postmenopausal bleeding. Mullerian congenital anomaly. Removal of foreign bodies. Undergoing the procedure to assess the endocervical canal, uterine cavity, and tubal ostia for infertility.

Exclusion Criteria:

* Patients with contra-indications of diagnostic hysteroscopy as:

Unable to exclude pregnancy Acute pelvic infection Active genital herpes Profuse bleeding at the time of the procedure. Any usage of analgesic agent on the day of the procedure. Failure of entry of the cervical canal requiring cervical dilatation. Any additional procedure during the procedure: polypectomy, biopsy and adhesiolysis.

Patient refusal to participate in the study.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-12 (Actual)

PRIMARY OUTCOMES:
Pain score | at time of hysteroscopy and 15 minutes after it
  using visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided